CLINICAL TRIAL: NCT00003214
Title: Randomized Trial on Chemosensitivity Testing in Advanced Primary Ovarian Carcinoma (Phase III)
Brief Title: Chemosensitivity Testing to Assign Treatment for Patients With Stage III or Stage IV Ovarian Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: SAKK 45/94; SWS-SAKK-45/94; EU-97036
Record Dates: First submitted 1999-11-01; First posted 2004-08-02 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Ovarian Cancer
Keywords: stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Cisplatin; Cyclophosphamide; Doxorubicin; Paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: in vitro sensitivity-directed chemotherapy
Drug: paclitaxel

SUMMARY:
RATIONALE: Chemosensitizers may increase the effectiveness of a chemotherapy drug by making tumor cells more sensitive to the drug.

PURPOSE: Randomized phase III trial to study the effectiveness of chemosensitivity testing to assign treatment for patients with stage III or stage IV ovarian cancer who have undergone surgery.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether the use of a chemosensitivity assay to assign treatment improves the time to progression and response rates of patients with stage III/IV ovarian cancer.

OUTLINE: This is a randomized study. Patients are stratified according to size of tumor after debulking surgery, stage, and Swiss Group for Clinical Cancer Research center where treatment is received. Within 14 days after patients undergo debulking surgery, they are randomized to one of two treatment arms. Arm I: Patients randomized to this arm receive one of six treatment regimens: Regimen A - cisplatin/cyclophosphamide Regimen B - cisplatin/cyclophosphamide/doxorubicin Regimen C - carboplatin Regimen D - carboplatin/cyclophosphamide Regimen E - cisplatin/paclitaxel Regimen F - carboplatin/paclitaxel Arm II: Patients who are randomized to this arm are assigned a treatment regimen based on a chemosensitivity assay of tumor specimens collected after debulking surgery. If no valid assay result is obtained, patients receive carboplatin/cyclophosphamide. Treatment is repeated every 3-4 weeks for a total of 6 courses. Up to 4 more courses may be administered if a partial response is demonstrated. Patients are followed every 3 months for the first 2 years and every 6 months thereafter.

PROJECTED ACCRUAL: Approximately 300 patients will be accrued for this study over 6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically/pathologically confirmed stage III and IV ovarian cancer Complete surgical staging and debulking including total abdominal hysterectomy, bilateral salpingo-oophorectomy, omentectomy, and biopsies of suspicious lesions (if feasible) required No low malignant potential histology without any invasive lesions in the peritoneum

PATIENT CHARACTERISTICS: Age: 80 and under Performance status: 0-3 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No disorder that would prevent the application of any protocol treatment

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Max Age: 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 1996-07; Primary Completion 2000-04 (Actual); Study Completion 2000-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: O.R. Kochli, MD, Study Chair — Frauenspital, Basel
Locations (10):
- Switzerland (10):
  - Kantonspital Aarau, Aarau
  - Frauenspital, Basel, Basel
  - Office of Walter Weber-Stadelman, Basel
  - University Hospital, Basel
  - Inselspital, Bern, Bern
  - Hopital Cantonal Universitaire de Geneva, Geneva
  - Istituto Oncologico della Svizzera Italiana, Lugano
  - Burgerspital, Solothurn, Solothurn
  - City Hospital Triemli, Zurich
  - Klinik Hirslanden, Zurich

REFERENCES:
- [Background] Koechli OR, Delaloye JF, Maibach R, et al.: Ovarian carcinoma FIGO II and IV - results of a randomized multicenter feasibility study with the ATP cell viability chemosensitivity assay. [Abstract] Proceedings of the American Society of Clinical Oncology 16: A-1326, 1997.
- [Result] Mariotta M, Perewusnyk G, Koechli OR, Little JB, von Knebel Doeberitz M, Mirimanoff RO, Rutz HP. Dexamethasone-induced enhancement of resistance to ionizing radiation and chemotherapeutic agents in human tumor cells. Strahlenther Onkol. 1999 Aug;175(8):392-6. doi: 10.1007/s000660050027. PMID 10481771